CLINICAL TRIAL: NCT06719440
Title: Impact of Reducing the Irradiation Volume on Survival, Toxicity, and Quality of Life in Patients With Glioblastoma Treated With Radiochemotherapy: a Prospective Multicenter Randomised Study
Brief Title: Achieving a Better Outcome Through Limiting the Glioblastoma Clinical Target Volume
Acronym: BELGICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KCE23-1426
Record Dates: First submitted 2024-11-15; First posted 2024-12-05 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; Radiotherapy Side Effect
MeSH Terms: conditions — Glioblastoma; Radiation Injuries | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: single blinded, randomized, parallel
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Radiation: Radiotherapy (CTV=15mm)
- Interventional arm (Experimental)
  Interventions: Radiation: Radiotherapy (CTV=10mm)

INTERVENTIONS:
Radiation: Radiotherapy (CTV=10mm) — Radiotherapy with reduced irradiation volume CTV=10mm
  Arms: Interventional arm
Radiation: Radiotherapy (CTV=15mm) — Radiotherapy with standard irradiation volume CTV=15mm
  Arms: Standard of Care

SUMMARY:
The objective of the BELGICA trial is to evaluate if radiotherapy could be given in a more focused manner in patients with glioblastoma in order to reduce side effects and improve quality of life.

The glioblastoma (GBM) is the most common and aggressive tumour originating from the brain, affecting approximately 600 patients per year in Belgium. The treatment consists in surgical resection of the tumour (when feasible), followed by a combination of radiotherapy and chemotherapy. Despite multimodal treatment (surgery, radiotherapy, and chemotherapy), the life expectancy of patients with GBM remains limited, with an average survival of 12-18 months and only 5% of patients surviving more than 5 years. In addition to limited survival, most patients with GBM experience impaired quality of life, both because of the disease and treatments.

Radiotherapy is a treatment where radiation is used to kill cancer cells. In GBM, radiotherapy is targeted at the tumour (or tumour bed if the tumour was resected) with a safety margin around it (the "Clinical Target Volume" or CTV) to account for potential microscopic spread of the tumour. The downside of this safety margin is that a substantial amount of brain tissue is irradiated, which can lead to treatment toxicity. Reducing the CTV margin would enable to decrease the volume of brain being irradiated and could thereby allow to reduce the side effects of brain irradiation.

The BELGICA trial (Achieving a BEtter outcome through Limiting the GlIoblastoma Clinical tArget volume) is a national multicentre trial which will evaluate if reducing the irradiation volume in glioblastoma is safe and allows for lowering side effects and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of giving informed consent
* Age >= 18 y.o.
* WHO performance status 0-2
* Newly diagnosed glioblastoma (Histologically proven glioblastoma per WHO 2021 classification based on biopsy or resection )
* Indication of chemoradiotherapy confirmed by multidisciplinary tumour board

Exclusion Criteria:

* Participation in a competing trial
* Known contraindication to undergo MRI scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From randomization to the end of the study
  Number of days from date of randomization to the date of death due to any cause

SECONDARY OUTCOMES:
Neurocognitive functioning | at baseline, 1 month after radiotherapy and at 1 year
  Hopkins verbal learning test revised; Trail Marking Test A & B; Controlled Oral Word Association Test
Radiation-induced toxicity | From enrollment until end of follow-up (2 years)
  Assessment of fatigue, headache, nausea, alopecia and radiatio dermatitis according to the CTCAE assessment score. Score ranges from Grade 1 to Grade 5, with higher grades resulting in more severe symptoms.
Health-related Quality of Life | From enrollment until end of follow-up (2 years)
  EQ-5D-5L; QLQ-C30; QLQ-BN20
Progression-free survival | From randomization until end of follow-up (2 years)
  Length of time during and after treatment for a disease, such as cancer, that a patient lives with the disease without it worsening
Pattern of recurrence | From randomization until end of follow-up (2 years)
  (in case of progression) Manner in which the tumor returns after a period of improvement or remission. It often involves tracking the frequency, timing, and location of the tumor's return
Anti-edema therapy | From randomization until end of follow-up (2 years)
  Recording of the needs of anti-edema therapy

OTHER OUTCOMES:
Normal tissue complication probability model (NTCP) | From enrollment until end of follow-up (2 years)
  To develop a normal tissue complication probability model (NTCP) for radiation-induced cognitive toxicity, based on clinical and dosimetric measures (e.g. radiation dose delivered to brain structures)

CONTACTS AND LOCATIONS:
Overall Officials: Dario Di Perri, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (23):
- Belgium (23):
  - Olv Azorg, Aalst
  - EpiCURA, Baudour
  - AZ Sint Jan, Bruges
  - Institut Jules Bordet, Brussels
  - UZ Brussel, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Ziekenhuis Oost-Limburg (ZOL), Genk
  - AZ Sint-Lucas, Ghent
  - UZ Gent, Ghent
  - Grand Hôpital de Charleroi, Gilly
  - JESSA Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - Chu Helora, La Louvière
  - UZ Leuven, Leuven
  - CHU Liège, Liège
  - AZ Sint Maarten, Mechelen
  - Hôpital André Vésale - HUmani, Montigny-le-Tilleul
  - CH Mouscron, Mouscron
  - CHU UCL Namur - Sainte Elisabeth, Namur
  - AZ Delta, Roeselare
  - Cliniques de l'Europe, Uccle
  - CHR Verviers, Verviers
  - ZAS Augustinus, Wilrijk

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT06719440/ICF_000.pdf